CLINICAL TRIAL: NCT06732752
Title: Prospective Validation of the New Trauma Score (NTS) for Superior Prediction of Mortality Compared to the Revised Trauma Score
Brief Title: Evaluating the New Trauma Score (NTS) for Improved Mortality Prediction
Acronym: NTS
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241210A; 009 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Trauma
Keywords: RTS
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective cohort study is to evaluate the predictive accuracy of the New Trauma Score (NTS), a modification of the Revised Trauma Score (RTS), in determining mortality outcomes among trauma patients admitted to the emergency department at Al-Kadhimiya Teaching Hospital, Iraq.

The main questions it aims to answer are:

Does the NTS provide a more accurate prediction of mortality than the RTS? Are there specific subgroups of trauma patients where the NTS demonstrates superior predictive utility compared to the RTS?

Participants will:

Be assessed using both the NTS and RTS upon admission to the emergency department.

Have their clinical outcomes, including mortality, tracked throughout their hospital stay.

DETAILED DESCRIPTION:
Trauma is increasingly being a cause of mortality globally. Every year, over 45 million people suffer moderate to severe disability as a result of trauma, making them the leading cause of mortality among persons aged 18 to 29. According to the World Health Organization (WHO), road traffic injuries caused 1.25 million deaths in 2014, and trauma is predicted to become the third biggest cause of disability globally by 2030. Accurate management and time are vital factors in the treatment of traumatic patients and play a main role in determining the outcome of trauma patients. Patients with serious traumatic injuries have a significantly lower likelihood of mortality or morbidity when treated at a designated trauma center.

Trauma scoring systems are simple to inform physicians of the severity of trauma in patients and help them decide the course of trauma management. They can be used in the field to determine whether to send a patient to a trauma center before they arrive at the hospital. When a trauma patient has just arrived at the emergency department (ED), they might also be utilized for clinical decision-making. Trauma scoring systems can be used in the emergency department to prepare the patient for surgery, to call on medical staff for trauma support, and to tell the patient's family of the severity of the patient's condition at an early stage. A scoring system must be accurate, reliable, and specific to predict trauma-related death.

As a result, trauma scores could be physiological, which detail changes in vital signs and state of awareness, such as the New Trauma Score (NTS) and Revised Trauma Score (RTS), which enable early clinical assessment of patients at admission. Anatomical, which describes the extent and number of anatomical lesions, such as the Abbreviated Injury Scale (AIS) and Injury Severity Score (ISS), allowing for later clinical assessment, including imaging after initial patient stabilization, surgery, and autopsy. combined, such as Trauma and Injury Severity Score (TRISS) and KTS, which incorporate RTS and ISS. The combined trauma ratings are especially useful in assessing the prognosis after trauma. Physiological NTS and combined KTS were developed primarily for their applicability in resource-constrained environments where advanced initial evaluation for anatomical lesions using computerized tomographic (CT) scans and magnetic resonance imaging (MRI) may not be available.

The New Trauma Score (NTS) is gaining popularity as an improved measure for predicting trauma mortality. It was created as a modification of the Revised Trauma Score (RTS) to enhance accuracy and usability. Compared to RTS, NTS includes extra measures such as oxygen saturation (SpO2) instead of respiratory rate, uses the actual Glasgow Coma Scale (GCS) score rather than coded values, and revise the systolic blood pressure interval used for the code value.These changes make the score more dynamic and suitable for a wider range of trauma settings.

Recent studies have validated the effectiveness of NTS. For instance, it demonstrated superior sensitivity in predicting mortality compared to the Kampala Trauma Score II (KTS II), though KTS II showed slightly higher specificity. NTS also performed well against other tools like MGAP and GAP, highlighting its balance between simplicity and precision. These features make it particularly useful in prehospital and emergency department triage systems, where rapid and reliable decisions are critical for patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients (including blunt, penetrating, and traumatic brain injury) admitted to the emergency department.
* Patients presenting with varying degrees of trauma (mild to severe).
* Patients (or their legal representatives) who provide informed consent to participate in the study.
* Trauma patients admitted to the emergency department.
* Patients who are assessed using both the Revised Trauma Score (RTS) and the New Trauma Score (NTS) upon admission to the emergency department.

Exclusion Criteria:

* Patients under 18 years old.
* Pregnant women, due to the potential complications and challenges in trauma assessment.
* Patients who refuse to give consent to participate in the study or whose legal guardians refuse on their behalf.
* Trauma patients transferred from other hospitals.
* Patients with incomplete medical records or missing key data required for trauma score calculation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consist of trauma patients admitted to the emergency department (ED) of Al-Kadhimiya Teaching Hospital over the study period. This will include both male and female patients of various age groups who present with trauma-related injuries.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7 days through discharge); Post-Discharge Follow-Up: Day 7, Day 30
  Mortality (death) during hospitalization
Accuracy Assessment of the New Trauma Score (NTS) | the first 6 hours after ER admission
  The New Trauma Score (NTS) ranges from 3 to 23. Higher scores indicate better physiological status and lower mortality risk.
Accuracy Assessment of the Revised Trauma Score (RTS) | the first 6 hours after ER admission
  The total RTS score ranges from 0 to approximately 12, with lower scores indicating more severe injuries and a higher risk of mortality.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Need for ICU Admission | Up to discharge, an average of 7 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.
Need for Surgical Intervention | Up to discharge, an average of 7 days
  need for surgical intervention during a trauma patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A. Hamdawi, Lecturer of general surgery, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manoochehry S, Vafabin M, Bitaraf S, Amiri A. A Comparison between the Ability of Revised Trauma Score and Kampala Trauma Score in Predicting Mortality; a Meta-Analysis. Arch Acad Emerg Med. 2019 Jan 15;7(1):e6. eCollection 2019 Winter. PMID 30847441
- [Background] Indurkar SK Sr, Ghormade PS, Akhade S, Sarma B. Use of the Trauma and Injury Severity Score (TRISS) as a Predictor of Patient Outcome in Cases of Trauma Presenting in the Trauma and Emergency Department of a Tertiary Care Institute. Cureus. 2023 Jun 14;15(6):e40410. doi: 10.7759/cureus.40410. eCollection 2023 Jun. PMID 37456404
- [Background] Mehmood A, Rowther AA, Kobusingye O, Ssenyonjo H, Zia N, Hyder AA. Delays in emergency department intervention for patients with traumatic brain injury in Uganda. Trauma Surg Acute Care Open. 2021 Aug 26;6(1):e000674. doi: 10.1136/tsaco-2021-000674. eCollection 2021. PMID 34527810
- [Background] MacKenzie EJ, Rivara FP, Jurkovich GJ, Nathens AB, Frey KP, Egleston BL, Salkever DS, Scharfstein DO. A national evaluation of the effect of trauma-center care on mortality. N Engl J Med. 2006 Jan 26;354(4):366-78. doi: 10.1056/NEJMsa052049. PMID 16436768
- [Background] Nirula R, Maier R, Moore E, Sperry J, Gentilello L. Scoop and run to the trauma center or stay and play at the local hospital: hospital transfer's effect on mortality. J Trauma. 2010 Sep;69(3):595-9; discussion 599-601. doi: 10.1097/TA.0b013e3181ee6e32. PMID 20838131
- [Background] Bachani AM, Peden M, Gururaj G, Norton R, Hyder AA. Road Traffic Injuries. In: Mock CN, Nugent R, Kobusingye O, Smith KR, editors. Injury Prevention and Environmental Health. 3rd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2017 Oct 27. Chapter 3. Available from http://www.ncbi.nlm.nih.gov/books/NBK525212/ PMID 30212112
- [Background] Byass P, de Courten M, Graham WJ, Laflamme L, McCaw-Binns A, Sankoh OA, Tollman SM, Zaba B. Reflections on the global burden of disease 2010 estimates. PLoS Med. 2013;10(7):e1001477. doi: 10.1371/journal.pmed.1001477. Epub 2013 Jul 2. PMID 23843748
- [Background] van Breugel JMM, Niemeyer MJS, Houwert RM, Groenwold RHH, Leenen LPH, van Wessem KJP. Global changes in mortality rates in polytrauma patients admitted to the ICU-a systematic review. World J Emerg Surg. 2020 Sep 30;15(1):55. doi: 10.1186/s13017-020-00330-3. PMID 32998744
- [Result] Damulira J, Muhumuza J, Kabuye U, Ssebaggala G, Wilson ML, Barnighausen T, Lule H. New Trauma Score versus Kampala Trauma Score II in predicting mortality following road traffic crash: a prospective multi-center cohort study. BMC Emerg Med. 2024 Jul 29;24(1):130. doi: 10.1186/s12873-024-01048-0. PMID 39075406
- [Result] Farzan N, Foroghi Ghomi SY, Mohammadi AR. A retrospective study on evaluating GAP, MGAP, RTS and ISS trauma scoring system for the prediction of mortality among multiple trauma patients. Ann Med Surg (Lond). 2022 Mar 28;76:103536. doi: 10.1016/j.amsu.2022.103536. eCollection 2022 Apr. PMID 35495411
- [Result] Chawda MN, Hildebrand F, Pape HC, Giannoudis PV. Predicting outcome after multiple trauma: which scoring system? Injury. 2004 Apr;35(4):347-58. doi: 10.1016/S0020-1383(03)00140-2. PMID 15037369
- [Result] Jeong JH, Park YJ, Kim DH, Kim TY, Kang C, Lee SH, Lee SB, Kim SC, Lim D. The new trauma score (NTS): a modification of the revised trauma score for better trauma mortality prediction. BMC Surg. 2017 Jul 3;17(1):77. doi: 10.1186/s12893-017-0272-4. PMID 28673278